CLINICAL TRIAL: NCT05348070
Title: Comparison of Inflammatory Parameters in Operated Ruptured and Non-ruptured Endometriomas
Brief Title: Comparison of Operated Ruptured and Non-ruptured Endometriomas
Acronym: RupturedOMA
Status: Completed | Type: Observational
Sponsor: EZH EAH (Other)
Responsible Party: Principal Investigator, MD. Ayşe Gülen Erturun, Principal Investigator, EZH EAH
Other Study IDs: 2021/76
Record Dates: First submitted 2022-01-25; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Endometrioma; Ruptured Endometrioma; Endometriosis Ovary
Keywords: endometrioma; rupture; endometriosis
MeSH Terms: conditions — Endometriosis; Rupture | interventions — Laparoscopy; Laparotomy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — all patients who were operated for endometrioma and had a histopathology report confirming the presence of endometrioma Surgical materials were biospecimens, which had a histopathology report confirming the presence of endometrioma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Operated Non-Ruptured Endometrioma Group: It consists of patients who were found to have endometrioma in their clinical follow-ups and decided to operate as a result of the evaluations. The patients were operated under elective conditions.
  Interventions: Procedure: Laparoscopy/Laparotomy
- Operated Ruptured Endometrioma Group: Rupture of endometrioma, which is a rare gynecological emergency. This group consists of endometrioma patients requiring urgent/subacute operation such as acute abdominal pain, hemodynamic instability, intra-abdominal bleeding. The patients were operated after completing the necessary preparations
  Interventions: Procedure: Laparoscopy/Laparotomy

INTERVENTIONS:
Procedure: Laparoscopy/Laparotomy — All patients included in the study were operated patients.

SUMMARY:
Ruptured endometrioma cases were compared with unruptured endometrioma cases.

DETAILED DESCRIPTION:
This study aims to compare the findings in patients who had surgery for ruptured endometrioma with the patients who had an unruptured endometrioma.

This study was conducted at Republic of Turkey Ministry of Health, Health Science University Etlik Zübeyde Hanım Gynecology Training and Research Hospital Infertility Clinic and all patients who were operated for endometrioma and had a histopathology report confirming the presence of endometrioma between January 2014 and December 2020 were included.

In this study, demographic characteristics, intraoperative findings, laboratory values and follow-up recommendations of two groups compared. The patients' age, presence of sexual activity and/or infertility, gravidity, parity, abortion, history of ectopic pregnancy, accompanying systemic disease, previous operations, drug use, and symptoms were recorded. Preoperative and postoperative complete blood count, Cancer antigen 125 (CA 125), Cancer antigen 19-9 (CA19-9), Cancer antigen 15-3 (CA 15-3), Carcinoembryonic antigen (CEA), alpha fetoprotein (AFP), anti mullerian hormone (AMH), fibrinogen, C-reactive protein (CRP) values of the patients were obtained. Patient files, operation notes and laboratory values of the electronic recording system database and the two groups were compared.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were operated on in Republic of Turkey Ministry of Health, Health Science University Etlik Zübeyde Hanım Gynecology Training and Research Hospital Infertility Clinic, whose histopathological diagnosis was confirmed as endometrioma, and who did not meet the exclusion criteria, were included in the study.

Exclusion Criteria:

* Patients who were operated with a prediagnosis of endometrioma and whose pathological diagnosis was different
* Patients with smoking, alcohol, substance abuse
* Patients receiving pelvic radiotherapy/chemotherapy
* Patients with suspected or confirmed malignancies

Ages: 16 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — The research was conducted on female patients.
Study Population: Patients who were operated on in Republic of Turkey Ministry of Health, Health Science University Etlik Zübeyde Hanım Gynecology Training and Research Hospital Infertility Clinic, whose histopathological diagnosis was confirmed as endometrioma. All patients were women of reproductive age with a pelvic mass.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Pre-interventional Comparison of inflammatory parameters | Blood samples were taken from the patients before the surgery
  Neutrophil/Lymphocyte ratio (NLR), Platelet/Lymphocyte ratio (PLR), Monocyte/Lymphocyte ratio (MLR) were compared between two groups in the preoperative period
Comparison of inflammatory parameters after surgery | Blood samples were taken from the patients in the first postoperative day.
  Neutrophil/Lymphocyte ratio (NLR), Platelet/Lymphocyte ratio (PLR), Monocyte/Lymphocyte ratio (MLR) were compared between two groups in the postoperative period
Pre-interventional Comparison of tumor markers | Blood samples were taken from the patients before the surgery
  Cancer antigens; CA125, CA19-9 and CA 15-3 were compared between two groups in the preoperative period
Comparison of tumor markers after surgery | Blood samples were taken from the patients after the surgery up to 24 weeks
  Cancer antigens; CA125, CA19-9 and CA 15-3 were compared between two groups in the postoperative period

SECONDARY OUTCOMES:
Sexual activity | Before surgery
  The existence of sexual activity in each study group was questioned.
Infertility | Before surgery
  The existence of infertility in each study group was questioned.

CONTACTS AND LOCATIONS:
Overall Officials: Berna Dilbaz, Prof., Study Director — Etlik Zübeyde Hanım Gynecology Training and Research Hospital Infertility Clinic's Chief
Locations (1):
- Republic of Turkey Ministry of Health, Health Science University Etlik Zübeyde Hanım Gynecology Training and Research Hospital Infertility Clinic, Ankara, Keçiören, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dai X, Jin C, Hu Y, Zhang Q, Yan X, Zhu F, Lin F. High CA-125 and CA19-9 levels in spontaneous ruptured ovarian endometriomas. Clin Chim Acta. 2015 Oct 23;450:362-5. doi: 10.1016/j.cca.2015.09.019. Epub 2015 Sep 25. PMID 26403090
- [Background] Huang YH, Liou JD, Hsieh CL, Shiau CS, Lo LM, Chang MY. Long-term follow-up of patients surgically treated for ruptured ovarian endometriotic cysts. Taiwan J Obstet Gynecol. 2011 Sep;50(3):306-11. doi: 10.1016/j.tjog.2010.05.002. PMID 22030044
- [Result] Tanaka K, Kobayashi Y, Dozono K, Shibuya H, Nishigaya Y, Momomura M, Matsumoto H, Iwashita M. Elevation of plasma D-dimer levels associated with rupture of ovarian endometriotic cysts. Taiwan J Obstet Gynecol. 2015 Jun;54(3):294-6. doi: 10.1016/j.tjog.2014.09.010. PMID 26166344